CLINICAL TRIAL: NCT03277404
Title: Effect of Smear Layer on Endodontic Outcome: A Randomized Controlled Trial
Brief Title: Effect of Smear Layer on Endodontic Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jyoti Rana
Record Dates: First submitted 2017-06-25; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-06

CONDITIONS: Apical Periodontitis
Keywords: EDTA; Postoperative pain; Pulp necrosis; Smear layer
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative; Dental Pulp Necrosis; Smear Layer | interventions — Therapeutic Irrigation; Edetic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smear Layer Positive (Experimental): Root canal treatment without smear layer removal: Root canal treatment and Irrigation with 1 ml of 2.5% sodium' hypochlorite for 1 min, followed by ultrasonic activation of 3 ml of 2.5% sodium hypochlorite for 1minute.
  Interventions: Procedure: Root canal treatment without smear layer removal
- Smear layer negative (Active Comparator): root canal treatment with smear layer removal:Root canal treatment and Irrigation with 1 mL of 17% EDTA solution and ultrasonic activation, followed by ultrasonic activation of 3 ml of 2.5% sodium hypochlorite for 1 minute.
  Interventions: Procedure: Root canal treatment with smear layer removal

INTERVENTIONS:
Procedure: Root canal treatment with smear layer removal — Canal were irrigated with Naocl and EDTA to remove smear layer
  Other Names: irrigation with EDTA
  Arms: Smear layer negative
Procedure: Root canal treatment without smear layer removal — only sodium hypochlorite was used for irrigation
  Other Names: irrigation with only NAOCL
  Arms: Smear Layer Positive

SUMMARY:
This study evaluated the effect of removal of smear layer on the success of primary root canal treatment.Patients requiring primary root canal treatment in mature mandibular first and second molars were allocated to either smear layer positive group and smear layer negative group.

DETAILED DESCRIPTION:
Patients requiring primary root canal treatment following the diagnosis of pulp necrosis in permanent mandibular first and second molars having radiographic evidence of periapical radiolucency (minimum size ≥ 2.0 × 2.0 mm) were included in the study. All patients were over 18 years of age and diagnosis of pulpal necrosis was confirmed by negative response to cold and electrical tests, and absence of bleeding on entering the pulp chamber. Patients with systemic illness, history of analgesic intake within past 7 days, antibiotics in the last 3months and patients who were pregnant were excluded from the study. Periodontally compromised teeth, previously accessed teeth, teeth that were not suitable for rubber dam isolation were also excluded from the study.

Subjects were allocated to one of the two study groups: smear layer positive group (only 2.5%NaOCl was used) - SP and smear layer negative group (17% EDTA+2.5%NaOCl was used) - SN. Using an equal proportion randomization allocation ratio, patients were assigned to the two groups using envelopes containing concealed assignment codes. It was ensured that neither the patient, nor the primary investigator was aware of the group till the time of final rinse.

After administration of local anesthesia, rubber dam isolation of the involved tooth was done. Caries was excavated and access cavity prepared using carbide burs in high speed handpiece with copious irrigation.Debridement of the pulp chamber was done and all canal orifices identified.Working length was obtained with the help of electronic apex locator and confirmed radiographically.Hand files number 10, 15 and 20 were used till working length (WL) to prepare a smooth reproducible glide path.Canal preparation was done with the help of rotary NiTi files. In both groups, 2.5% sodium hypochlorite was used as irrigant after each instrument. All the irrigation procedures were performed using a 27 gauge side vented needle. After root canal instrumentation, 17% Ethylenediaminetetraacetic acid (EDTA) solution was also used to remove smear layer in smear layer negative group, while teeth in smear layer positive group was simply rinsed with 2.5% sodium hypochlorite. In both the groups ultrasonic activation of irrigant was done. An inter-appointment dressing of calcium hydroxide was given. The access cavity was then restored with intermediate restorative material (Dental Products of India).

Patients were prescribed Ibuprofen 400mg with the instructions to take one tablet every 8 hours in the event of pain.Patients were asked to record the severity of pain using 10 cm VAS scale with 0 depicting no pain and 10 depicting maximum pain imaginable. Patients were asked to make a mark on the line that represented their level of perceived pain every 24hrs for 7 days following intervention.

One week later, patients returned with the completed questionnaires.

At the same appointment the intracanal dressing was removed with H-files and copious irrigation with 2.5% NaOCl in both the groups.

17% EDTA solution was used to remove smear layer in smear layer negative group, followed by 2.5% NaOCl while teeth in smear layer positive group were simply rinsed with 2.5% sodium hypochlorite.

Ultrasonic activation of irrigant was done and canals were obturated with the GuttaPercha and Zinc Oxide-Eugenol based sealer in both the groups. After obturation, the cavity was restored permanently.Immediate post-operative radiograph was then taken using preset exposure parameters.Follow up clinical and radiographic examination was carried out every 3 months, till a 12 month period. The data gathered was analyzed using suitable statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent mandibular first and second molars requiring primary root canal treatment
* Diagnosis of pulpal necrosis, as confirmed by negative response to cold and electrical tests; and absence of bleeding on entering the pulp chamber
* Radiographic evidence of periapical radiolucency (minimum size ≥ 2.0 × 2.0 mm)
* Patient's age more than 18 years

Exclusion Criteria:

* Patients who do not provide consent for participation in the study
* Age <18 years
* Positive history of antibiotic use within past one month of the treatment
* Patients who are pregnant, diabetic, immunocompromised, had serious medical illness or required antibiotic premedication
* Patients with pockets ≥4mm or having marginal or furcal bone loss due to periodontitis
* Teeth that are not suitable for rubber dam isolation
* Previously accessed teeth and/or with procedural errors
* Unrestorable tooth, fractured/ perforated roots, inflammatory root resorption

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Radiographic success | every 3 months till 12 month period
  Size of apical radiolucency were scored according to PAI scores and PAI score less than 3 were considered as success
Clinical success | till 12 months
  Presence or absence of any clinical symptoms such as pain,tenderness, sinus tract and swelling

SECONDARY OUTCOMES:
Pain intensity | Patients were asked to make a mark on the line that represented their level of perceived pain every 24hrs for7 days following intervention
  Pain intensity before and after treatment. Intensity of pain was recorded using 10 cm VAS scale with 0 depicting no pain and 10 depicting maximum pain imaginable.

IPD SHARING:
Plan to Share IPD: No